CLINICAL TRIAL: NCT01289821
Title: An Uncontrolled, Open-label, Phase II Study in Subjects With Metastatic Adenocarcinoma of the Colon or Rectum Who Are Receiving First Line Chemotherapy With mFOLFOX6 (Oxaliplatin/ Folinic Acid/5-fluorouracil [5-FU]) in Combination With Regorafenib
Brief Title: First Line Treatment of Metastatic Colorectal Cancer With mFOLFOX6 in Combination With Regorafenib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11728; 2010-020121-41 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib + oxaliplatin/folinic acid/5-FU (mFOLFOX6) (Experimental): On Day 1, participants received 85 mg/m^2 oxaliplatin as a 2-hour intravenous (IV) infusion and folinic acid (either 400 mg/m^2 D/L-folinic acid or 200 mg/m^2 L-folinic acid) as a 2-hour IV infusion. Once the initial infusion was completed, participants received 5-FU 400 mg/m^2 IV bolus injection immediately followed by a 5-FU 2400 mg/m^2 IV infusion for 46 hours. The next cycle of mFOLFOX6 was administered on Day 15 to 17. Participants received Regorafenib (Stivarga, BAY73-4506) 160 mg orally (po) once daily (qd) on Days 4 to 10 and Days 18 to 24. One cycle comprised 28 days.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-FU (mFOLFOX6)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Subjects will receive regorafenib 160 mg od on days 4 to 10 and days 18 to 24 as four 40 mg coprecipitate tablets. In case of administration as a single agent during the study, regorafenib will be administered 160 mg od for 3 weeks on/1 week off. Each cycle consists of 28 days.
Drug: Oxaliplatin — On day 1 and day 15 of each cycle, participants will receive 85 mg/m^2 oxaliplatin as a 2 hour i.v. infusion.
Drug: Folinic acid — On day 1 and day 15 of each cycle, participants will receive folinic acid (either 400 mg/m^2 D/L-folinic acid or 200 mg/m^2 L-folinic acid) as a 2 hour i.v. infusion.
Drug: 5-FU (mFOLFOX6) — Participants will receive a 400 mg/m^2 5 FU i.v. bolus injection immediately followed by a 2400 mg/m^2 5 FU 46 hour i.v. infusion.

SUMMARY:
This is a study to evaluate the efficacy (effectiveness) and the safety of regorafenib when given in combination with chemotherapy mFOLFOX6 as first line therapy in patients with metastatic colorectal cancer (CRC). mFOLFOX6 is an approved chemotherapy. Regorafenib is an oral (i.e. taken by mouth) multi-targeted kinase inhibitor. A kinase inhibitor targets certain key proteins that are essential for the survival of the cancer cell. By specifically targeting these proteins, regorafenib may stop cancer growth. The growth of the tumor may be decreased by preventing these specific proteins from functioning.

The primary endpoint (the most meaningful result to be tracked) of this study is based on the rate of response, i.e. the disease getting smaller. The aim is to show that the therapy of colorectal cancer with mFOLFOX6 in combination with regorafenib improves the response rate observed for the standard therapy only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years
* Histological or cytological documentation of adenocarcinoma of the colon or rectum
* Suitable to receive mFOLFOX6 regimen as first line metastatic treatment
* At least 1 measurable lesion as per RECIST version 1.1
* Unresectable or unlikely becoming resectable metastatic disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 3 months
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Prior systemic anticancer therapy for metastatic colorectal cancer (CRC). Adjuvant chemotherapy for CRC (Stage I, II, III) is permitted, if the adjuvant therapy ended > 6 months before screening and recurrent disease was documented.
* Prior treatment with antivascular endothelial growth factor (anti-VEGF) agents and any signal transduction inhibitors (STIs)
* Uncontrolled hypertension
* Subjects with symptoms, signs, or history of brain metastases
* Any hemorrhage or bleeding event ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 within 4 weeks of start of study treatment
* Sensory neuropathy (> CTCAE Grade 1), unresolved toxicity > CTCAE Grade 1 attributed to any prior therapy/procedure excluding alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Chicago, Illinois, United States
- Australia (2):
  - Concord, New South Wales
  - Woodville South, South Australia
- Belgium (3):
  - Bruxelles - Brussel
  - Edegem
  - Leuven
- Germany (4):
  - Stuttgart, Baden-Wurttemberg
  - Oldenburg, Lower Saxony
  - Herne, North Rhine-Westphalia
  - Dresden, Saxony
- Italy (3):
  - Napoli, Campania
  - Genoa, Liguria
  - Ancona, The Marches
- Spain (3):
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Madrid, Madrid
- United Kingdom (2):
  - Manchester, Manchester
  - Glasgow

REFERENCES:
- [Result] Schultheis B, Folprecht G, Kuhlmann J, Ehrenberg R, Hacker UT, Kohne CH, Kornacker M, Boix O, Lettieri J, Krauss J, Fischer R, Hamann S, Strumberg D, Mross KB. Regorafenib in combination with FOLFOX or FOLFIRI as first- or second-line treatment of colorectal cancer: results of a multicenter, phase Ib study. Ann Oncol. 2013 Jun;24(6):1560-7. doi: 10.1093/annonc/mdt056. Epub 2013 Mar 13. PMID 23493136
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female participants with histological or cytological documentation of adenocarcinoma of the colon or rectum that was unresectable or unlikely of becomining resectable, who were at least 18 years of age and were suitable to receive mFOLFOX6 regimen as first line treatment could participate in this study at 16 centers in 7 countries.
Pre-assignment Details: Of 66 enrolled participants, 54 received study medication, 4 withdrew consent during screening, and 8 were screen failures due to no measurable lesion, not suitable to receive mFOLFOX as 1st line regimen (2), uncontrolled hypertension, symptoms/signs/history of brain metastases, glomerular filtration rate too low (2), and protein in spot urine
Period: Treatment Period
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Started | 54
Participants Received Regorafenib | 54
Completed | 0
Not Completed | 54
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Adverse Event | 4
Not completed — Radiological Progression | 43
Not completed — Clinical Progression | 2
Not completed — Therapeutic procedure required | 1
Period: Safety Follow-up Period
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Started | 54
Completed | 49
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3
Not completed — Unspecified reason | 1
Period: Survival Follow-up Period
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Started | 52
Completed | 34 (34 participants died and completed survival follow-up period.)
Not Completed | 18
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Clinical endpoint reached | 16

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 54
Age, Customized [Number; unit: Participants]
  < 65 years | 33
  65 - 75 years | 18
  > 75 years | 3
Sex/Gender, Customized [Number; unit: Paricipants]
  Female | 26
  Male | 28
Caucasian [Number; unit: Participants] | 54
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at study entry [Number; unit: Participants] — The ECOG PS required for the study was 0 (fully active) or 1 (restricted in physically strenous activity but ambulatory and able to carry out work of a light or sedentary nature)
  Participants
    0 | 35
    1 | 19
Stage at initial diagnosis [Number; unit: Participants] — The TNM Classification of Malignant Tumors (TNM) is a cancer staging system that describes the extent of a person's cancer. T describes the size of the original (primary) tumor and whether it has invaded nearby tissue, N describes nearby (regional) lymph nodes that are involved, M describes distant metastasis. For colon carcinoma, this is translated into stages I-IV. Stages II-IV can be further subdivided in subgroups (eg, A,B, or C).
  Participants
    I | 1
    IIA | 5
    IIIB | 3
    IIIC | 4
    IV | 41

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR)
Description: OR was defined as the best tumor response (confirmed complete response [CR] or partial response [PR]) observed by MRI or CT scan assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1. CR and PR were confirmed not earlier than 4 weeks following the initial detection of response. CR = Disappearance of all clinical and radiological evidence of tumor (both target and no-target). Any pathological lymph nodes (whether target or non target) must have a reduction in short axis to < 10 mm. PR = At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing nontarget lesions and no appearance of new lesions.
Time Frame: From start of treatment until 30 days after termination of study medication, an average of 47 weeks. Assessed every 8 weeks.
Population: Primary analysis set (PAS, N=41) was a subset of the PPS and included the first 41 subjects, who were assigned to treatment
Measure: Number; unit: Proportion of participants
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 41
Proportion of participants | 0.4390
Statistical Analysis 1: Comparison: Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6); Null hypothesis: "True probability p of objective tumor response does not exceed p0, p0=0.4." H0: p<=0.4 One-sided type I error probability of alpha=10%; Test type: Superiority or Other; p = 0.36, One-sample exact binomial test; Percentage of Participants = 43.90, 80% CI 2-sided [33.19 to 55.09]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated as the time from first date of receiving study treatment to date of death due to any cause. Participants alive at the time of analysis were censored at their last date of follow-up.
Time Frame: From start of treatment until 30 days after the last dose of study treatment, assessed by every 8 weeks
Population: Full analysis set (FAS, N=54) included all subjects who received treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 54
Days | 772 [646 to 1089]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as time from the date of start of study treatment to the date of first observed disease progression (radiological according to central assessment or clinical), or death due to any cause, if death occurred before progression was documented. PFS for participants without disease progression or death at the date of database cutoff were right-censored at the last date of tumor assessment. Participants who had no tumor evaluation after baseline and no clinical progression post baseline and who did not die were censored at Day 1 in the analysis. PD = At least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non target lesions or the appearance of one or more new lesions will also constitute PD.
Time Frame: From start of treatment until 30 days after the last dose of study treatment, assessed by every 8 weeks
Population: Full analysis set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 54
Days | 258 [222 to 334]

4. Secondary Outcome: Disease Control (DC)
Description: DC was defined as the proportion of participants who had a best response rating of CR, PR, or stable disease (SD) according to RECIST criteria that was achieved during treatment or within 30 days after termination of study treatment. CR and PR were confirmed not earlier than 4 weeks following the initial detection of response. A minimum of 8 weeks (allowing a minus 7-day time window) between start of study treatment and the first follow-up tumor assessment with SD as response was required to assign SD as best overall response.
Time Frame: From start of treatment until 30 days after the last dose of study treatment, assessed by every 8 weeks
Population: PAS
Measure: Number; unit: Proportion of participants
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 41
Proportion of participants | 0.8537

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documented objective response of PR or CR, whichever was noted earlier, to first subsequent disease progression or death (if death occurred before progression was documented). DOR was defined for responders only (that is, subjects with CR or PR). DOR for subjects without disease progression or death before progression was right censored at the date of their last tumor assessment.
Time Frame: From start of treatment until 30 days after the last dose of study treatment, assessed by every 8 weeks
Population: Per protocol set (PPS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 20
Days | 257 [176 to 349]

6. Secondary Outcome: Duration of Stable Disease (DOSD)
Description: DOSD was only evaluated in participants failing to achieve a best response of CR or PR, but who achieved SD. DOSR was defined as the time (in days) from date of start of study treatment to the date at which disease progression or death (if death occurred before progression was first documented). The date the tumor scan was performed was used for this calculation. DOSD for participants without disease progression or death before progression at the time of analysis were censored at the date of their last tumor assessment.
Time Frame: From start of treatment until 30 days after the last dose of study treatment, assessed by every 8 weeks
Population: Per protocol set (PPS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Number analyzed (Participants) | 22
Days | 231 [167 to 259]

ADVERSE EVENTS:
Time Frame: From start of study treatment until 4 weeks following the last dose of study treatment.
Description: Of 54 treated subjects, 53 subjects were valid for safety population. One subject was excluded from the SAF. The reason for the exclusion "never received regorafenib" is only enumerated once, under the reasons for exclusion from the SAF.
Groups:
- Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6): On Day 1, participants received 85 mg/m2 oxaliplatin as a 2-hour intravenous (IV) infusion and folinic acid (either 400 mg/m2 D/L folinic acid or 200 mg/m2 L-folinic acid) as a 2-hour IV infusion. Once the initial infusion was completed, participants received 5-FU 400 mg/m2 IV bolus injection immediately followed by a 5-FU 2400 mg/m2 IV infusion for 46 hours. The next cycle of mFOLFOX6 was administered on Day 15 to 17. Participants received Regorafenib (Stivarga, BAY73-4506) 160 mg orally (po) once daily (qd) on Days 4 to 10 and Days 18 to 24. One cycle comprised 28 days.
Arm/Group | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6)
Serious Adverse Events (participants affected / at risk) | 25/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6) (N=53)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Infusion related reaction (General disorders) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 7 (9)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib + Oxaliplatin/Folinic Acid/5-FU (mFOLFOX6) (N=53)
Anemia (Blood and lymphatic system disorders) | 12 (25)
Conduction disorder (Cardiac disorders) | 4 (8)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 28 (47)
Constipation (Gastrointestinal disorders) | 17 (26)
Diarrhea (Gastrointestinal disorders) | 37 (124)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Mucositis oral (Gastrointestinal disorders) | 24 (65)
Nausea (Gastrointestinal disorders) | 28 (70)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 16 (29)
Fatigue (General disorders) | 34 (92)
Fever (General disorders) | 10 (18)
Infusion related reaction (General disorders) | 3 (7)
Injection site reaction (General disorders) | 4 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (4)
Pain (General disorders) | 13 (15)
Alanine aminotransferase increased (Investigations) | 10 (27)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 12 (29)
Blood bilirubin increased (Investigations) | 9 (15)
GGT increased (Investigations) | 8 (17)
Lipase increased (Investigations) | 14 (19)
Neutrophil count decreased (Investigations) | 35 (88)
Investigations - Other, specify (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 25 (61)
Serum amylase increased (Investigations) | 5 (8)
White blood cell decreased (Investigations) | 6 (8)
Weight loss (Investigations) | 5 (7)
Allergic reaction (Immune system disorders) | 5 (5)
Catheter related infection (Infections and infestations) | 3 (5)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4)
Paronychia (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 6 (10)
Urinary tract infection (Infections and infestations) | 5 (7)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 21 (41)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (7)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (35)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (15)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Dizziness (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 16 (18)
Dysesthesia (Nervous system disorders) | 7 (14)
Headache (Nervous system disorders) | 8 (15)
Lethargy (Nervous system disorders) | 10 (29)
Paresthesia (Nervous system disorders) | 28 (71)
Peripheral sensory neuropathy (Nervous system disorders) | 24 (47)
Somnolence (Nervous system disorders) | 3 (4)
Conjunctivitis (Eye disorders) | 3 (4)
Eye disorders - Other, specify (Eye disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 12 (29)
Hematuria (Renal and urinary disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (5)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (47)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (10)
Flushing (Vascular disorders) | 5 (8)
Hypotension (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 30 (134)
Phlebitis (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI has to submit a draft manuscript of the publication or abstract to Bayer for review and approval at least 60 days before submission. Possible discrepancies will be discussed to find solution which satifies both parties. Bayer may delay publication for up to three months after analyzing the results.